CLINICAL TRIAL: NCT06708273
Title: Effect of Constraint Induced Movement Therapy on Burned Dominant Hand Function
Acronym: CIMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Elbadri Farouk Ahmed, Demonstrator, Cairo University
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P.T.REC/012/005218
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Effect of Constraint Induced Movement Therapy on Burned Dominant Hand Function; Hand Burn
Keywords: Hand function - CIMT - Constraint - Dominant; hand; function; constraint induced movement therapy; burn
MeSH Terms: conditions — Burns | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 received constraint induced movement therapy + traditional treatment (Experimental): group 1 received constraint induced movement therapy + traditional treatment we will constraint affected hand and enforce patient to use affected side
  Interventions: Other: Constraint induced movement therapy; Other: Positioning - stretching
- traditional treatment for hand burn positioning - RANGE OF MOTION (Active Comparator): traditional treatment for hand burn positioning - RANGE OF MOTION
  Interventions: Other: Positioning - stretching

INTERVENTIONS:
Other: Constraint induced movement therapy — Constraint the sound side and encourage movement of the burned side
  Other Names: CIMT
  Arms: group 1 received constraint induced movement therapy + traditional treatment
Other: Positioning - stretching — Position hand in functional hand position - stretching against deformity position
Other: constraint induced movement therapy — constraining sound hand to enforce patient to use affected burned dominant hand
  Arms: group 1 received constraint induced movement therapy + traditional treatment

SUMMARY:
Effect of constraint induced movement therapy on burned dominant hand function

DETAILED DESCRIPTION:
Effect of constraint induced movement therapy on burned dominant hand function

We investigate the Effect of constraint induced movement therapy on burned dominant hand function by using various measurement tools :

* Hand grip strength by Hand held dynamometer
* Metacarpophalangeal joint flexion (MCP) by goniometer
* Function by michgan hand questionnaire A randomised controlled trial (2 groups) First group will receive constraint induced movement therapy (glove mitt) on sound hand .

Second group will receive the traditional treatment ( stretching - positioning ) We do the assessment before treatment and (4-8) after the start of treatment process.

ELIGIBILITY:
Inclusion Criteria:

* Age of patient 20 to 35
* both male and female
* suffer from dorsal hand dominant burn healed spontaneously or by graft
* TBSA less than 20%
* All patient active before injury.

Exclusion Criteria:

* patient with fracture
* patient with crush injuries
* patient with contralateral hand burn
* Patient with cardiovascular injury

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2024-05-22 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
Hand grip strength | 8 weeks for each case
  Strength measured by hand held dynamometer
Metacarpophalangeal joint flexion | 8 weeks for each case
  Range of motion by goinometer
Hand function | 8 weeks for each case
  By arabic version of michgan hand qurstionaire

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided